CLINICAL TRIAL: NCT05572775
Title: Post-surgical Chronic Pain After Retroperitoneal Laparoscopic Living Kidney Donor in Cipto Mangunkusumo Hospital: Comparison Analysis of Brief Pain Inventory (BPI) in Erector Spinae Plane (ESP) Block VS Quadratus Lumborum (QL) Block
Brief Title: Post-surgical Chronic Pain After Retroperitoneal Laparoscopic Living Kidney Donor
Status: Completed | Type: Observational
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Indonesia University
Other Study IDs: Chronic Post-op Pain Donor
Record Dates: First submitted 2022-09-26; First posted 2022-10-10 (Actual); Last update posted 2023-09-07 (Actual); Status verified 2023-09

CONDITIONS: Chronic Post Operative Pain; Kidney Transplant; Complications; Anesthesia Regional; Laparoscopy
MeSH Terms: conditions — Pain, Postoperative | interventions — Dental Occlusion; Parapsychology

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Chronic post-surgical pain: Living kidney donor with the incidence of chronic post-surgical pain
  Interventions: Procedure: Quadratus lumborum (QL) block; Procedure: Erector Spinae Plane (ESP) Block
- Non-Chronic Post-surgical pain: Living kidney donor without the incidence of chronic post-surgical pain
  Interventions: Procedure: Quadratus lumborum (QL) block; Procedure: Erector Spinae Plane (ESP) Block

INTERVENTIONS:
Procedure: Quadratus lumborum (QL) block — bilateral anterior subcostal quadratus lumborum block
Procedure: Erector Spinae Plane (ESP) Block — bilateral erector spinae plane block

SUMMARY:
This study aimed to determine the relationship between the quadratus lumborum and erector spinae plane block technique and the incidence and severity of chronic post-surgical pain in accordance with Brief Pain Inventory Score (BPI) in retroperitoneal laparoscopic living kidney donor surgery

DETAILED DESCRIPTION:
A minimum of 130 subjects will be recruited and divided into two groups (65 QL block, 65 ESP block). The researcher will use the Brief Pain Inventory (BPI) score to assess the incidence and severity of chronic pain of the living kidney donor who has undergone retroperitoneal laparoscopy with QL or ESP block technique

ELIGIBILITY:
Inclusion Criteria:

* Patient 18-65 years old
* Patient with ASA physical status assessment 1-3
* All patient who have undergone living kidney donor with retroperitoneal laparoscopy at RSUPN Dr. Cipto Mangunkusumo (3 months postoperative)
* The patient and/ or the family are willing to be interviewed about the patient's previous medical history and agree to be the subject of the study.

Exclusion Criteria:

* Patient who have already known the cause of the chronic pain they had
* Patient who have history of major surgery after the donor surgery
* Patient died during the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population is all living kidney donor patients with retroperitoneal laparoscopy technique and performed QL or ESP block technique at RSUPN Dr. Cipto Mangunkusumo
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Chronic post-surgical pain | 3 months after surgery
  the correlation between QL and ESP block technique and the incidence of chronic post-surgical pain

SECONDARY OUTCOMES:
The incidence of chronic post-surgical pain | 3 months after surgery
  the incidence of patients with chronic post-surgical pain 3 months after surgery
The severity of chronic post-surgical pain Brief Pain Inventory (BPI) | 3 months after surgery
  the severity of chronic post-surgical pain 3 months after surgery. Assessed in The Brief Pain Inventory (BPI) short version. Zero (0) represent no pain and Ten (10) represent pain as bad as you can imagine.
Impact of chronic post-surgical pain on the daily activities (pain interferences) | 3 months after surgery
  Impact of chronic post-surgical pain on daily activities (pain interferences). Assessed using The Brief Pain Inventory (BPI), described in 0 (zero) does not interfere and 10 (ten) completely interferes daily activities.

CONTACTS AND LOCATIONS:
Locations (1):
- Cipto Mangunkusumo Hospital, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No